CLINICAL TRIAL: NCT04915001
Title: An Investigation on the Role of Emergency Departments in Combatting Against COVID-19 in Zhejiang Province
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Hospital (Other); Zhejiang Provincial People's Hospital (Other); Zhejiang Litongde Hospital (Unknown); Zhejiang University (Other); Sir Run Run Shaw Hospital (Other); The Fourth Affiliated Hospital of Zhejiang University School of Medicine (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Zhejiang Traditional Chinese Medicine Hospital (Unknown); The Third Affiliated Hospital of Zhejiang University of Traditional Chinese Medicine (Unknown); The 90th and Third Hospital of the Joint Logistics Support Force of the Chinese People's Liberation Army (Unknown); The 72nd Group Army Hospital of the Chinese People's Liberation Army (Unknown); Zhejiang Provincial Hospital of the Chinese People's Armed Police Force (Unknown); First People's Hospital of Hangzhou (Other); The Third People's Hospital of Hangzhou (Other); Red Cross Hospital, Hangzhou, China (Other); Hangzhou Traditional Chinese Medicine Hospital (Unknown); The Affiliated Hospital of Hangzhou Normal University (Other); Hangzhou Dajiangdong Hospital (Unknown); The First People's Hospital of Xiaoshan District (Unknown); The Second People's Hospital of Yuhang District (Unknown); The Third People's Hospital of Yuhang District (Unknown); Yuhang Hospital of Traditional Chinese Medicine (Unknown); The First People's Hospital of Fuyang District (Unknown); Fuyang District Traditional Chinese Medicine Hospital (Unknown); Lin'an People's Hospital (Unknown); Lin'an Traditional Chinese Medicine Hospital (Unknown); The First People's Hospital of Tonglu County (Unknown); Tonglu Hospital of Traditional Chinese Medicine (Unknown); The First People's Hospital of Chun'an County (Unknown); Chun'an County Hospital of Traditional Chinese Medicine (Unknown); The First People's Hospital of Jiande City (Unknown); Jiande City Hospital of Traditional Chinese Medicine (Unknown); The First People's Hospital of Huzhou (Other); Huizhou Municipal Central Hospital (Other); Huzhou Traditional Chinese Medicine Hospital (Unknown); Huzhou Third People's Hospital (Other); People's Hospital of Wuxing District, Huzhou City (Unknown); People's Hospital of Nanxun District, Huzhou City (Unknown); Anji County People's Hospital (Unknown); The Third People's Hospital of Anji County (Unknown); Deqing County People's Hospital (Unknown); Changxing People's Hospital (Other); Changxing County Hospital of Traditional Chinese Medicine (Unknown); Affiliated Hospital of Jiaxing University (Other); The Second Affiliated Hospital of Jiaxing University (Other); Jiaxing Traditional Chinese Medicine Hospital (Unknown); Haining People's Hospital (Unknown); Haining Traditional Chinese Medicine Hospital (Unknown); The First People's Hospital of Tongxiang City (Unknown); Haiyan County People's Hospital (Unknown); The First People's Hospital of Jiashan County (Unknown); Jiashan County Hospital of Traditional Chinese Medicine (Unknown); Zhejiang Xin'an International Hospital (Unknown); Jinhua Central Hospital (Other); Jinhua City People's Hospital (Unknown); Jinhua Traditional Chinese Medicine Hospital (Unknown); Yongkang Traditional Chinese Medicine Hospital (Unknown); Pujiang County People's Hospital (Unknown); Pujiang County Hospital of Traditional Chinese Medicine (Unknown); The First People's Hospital of Wucheng District, Jinhua City (Unknown); People's Hospital of Wucheng District, Jinhua City (Unknown); Second People's Hospital of Jindong District, Jinhua City (Unknown); Yiwu Central Hospital (Other); Dongyang People's Hospital (Other); Dongyang Traditional Chinese Medicine Hospital (Unknown); Lanxi People's Hospital (Other); Pan'an County People's Hospital (Unknown); Lanxi Traditional Chinese Medicine Hospital (Unknown); Hangzhou Medical College (Other); The First People's Hospital of Wuyi County (Unknown); The Central Hospital of Lishui City (Other); Lishui Traditional Chinese Medicine Hospital (Unknown); Liandu District People's Hospital (Unknown); Longquan People's Hospital (Unknown); Jinyun County People's Hospital (Unknown); Jingning County People's Hospital (Unknown); Qingtian County People's Hospital (Unknown); Qingyuan People's Hospital (Other); Songyang County People's Hospital (Unknown); Songyang County Hospital of Traditional Chinese Medicine (Unknown); Suichang County People's Hospital (Unknown); Yunhe County People's Hospital (Unknown); Ningbo No.2 Hospital (Other); Ningbo No. 1 Hospital (Other); Ningbo Third Hospital (Unknown); Li Huili Hospital, Ningbo Medical Center (Unknown); Ningbo Traditional Chinese Medicine Hospital (Unknown); Ningbo Ninth Hospital (Unknown); People's Hospital of Beilun District, Ningbo City (Unknown); Ningbo Yinzhou People's Hospital (Unknown); The Second Hospital of Yinzhou District, Ningbo City (Unknown); The Second Hospital of Haishu District, Ningbo City (Unknown); People's Hospital of Zhenhai District, Ningbo City (Unknown); People's Hospital of Fenghua District, Ningbo City (Unknown); Mingzhou Hospital of Zhejiang University (Unknown); Cixi City People's Hospital (Unknown); Ninghai County First Hospital (Unknown); Xiangshan County First People's Hospital Medical and Health Group (Unknown); People's Hospital of Quzhou (Other); Quzhou Second People's Hospital (Unknown); Zhejiang Quhua Hospital (Other); Quzhou Traditional Chinese Medicine Hospital (Unknown); People's Hospital of Kecheng District, Quzhou City (Unknown); Jiangshan City People's Hospital (Unknown); Jiangshan Traditional Chinese Medicine Hospital (Unknown); Jiangshan Beilin Hospital (Unknown); Kaihua County People's Hospital (Unknown); Kaihua County Hospital of Traditional Chinese Medicine (Unknown); Changshan County People's Hospital (Unknown); Longyou County People's Hospital (Unknown); Longyou County Hospital of Traditional Chinese Medicine (Unknown); Shaoxing People's Hospital (Other); Shaoxing Second Hospital (Other); Shaoxing Traditional Chinese Medicine Hospital (Unknown); Shangyu People's Hospital of Shaoxing City (Unknown); Shangyu Hospital of Traditional Chinese Medicine, Shaoxing City (Unknown); Traditional Chinese Medicine Hospital of Keqiao District, Shaoxing City (Unknown); Zhuji City People's Hospital (Unknown); Zhuji City Hospital of Traditional Chinese Medicine (Unknown); Shengzhou Traditional Chinese Medicine Hospital (Unknown); Xinchang County People's Hospital (Unknown); Taizhou Hospital (Other); Taizhou Enze Medical Center Group (Other); Taizhou First People's Hospital (Other); Taizhou Hospital of Traditional Chinese Medicine (Other Government); First People's Hospital of Linhai City (Unknown); Second People's Hospital of Linhai City (Unknown); Affiliated Wenling Hospital of Wenzhou Medical University (Other); Wenling Traditional Chinese Medicine Hospital (Unknown); Yuhuan City People's Hospital (Unknown); Sanmen County People's Hospital (Unknown); Tiantai County People's Hospital (Unknown); Xianju County People's Hospital (Unknown); Wenzhou Central Hospital (Other); Wenzhou People's Hospital (Other); Wenzhou Traditional Chinese Medicine Hospital (Unknown); Wenzhou Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); Lucheng District People's Hospital of Wenzhou City (Unknown); The First People's Hospital of Longwan District, Wenzhou City (Unknown); Wenzhou Longwan District Integrated Traditional Chinese and Western Medicine Hospital (Unknown); Wenzhou Ouhai District People's Hospital (Unknown); The Third People's Hospital of Ouhai District, Wenzhou City (Unknown); Wenzhou Ouhai District Hospital of Integrated Traditional Chinese and Western Medicine (Unknown); Wenzhou Dongtou District People's Hospital (Unknown); Affiliated Yueqing Hospital of Wenzhou Medical University (Other); The Second People's Hospital of Yueqing City (Unknown); The Third People's Hospital of Yueqing City (Unknown); The Fifth People's Hospital of Yueqing City (Unknown); Yueqing Traditional Chinese Medicine Hospital (Unknown); The Third Affiliated Hospital of Wenzhou Medical University (Other); Ruian City Hospital of Traditional Chinese Medicine (Unknown); Longgang People's Hospital (Unknown); Cangnan County People's Hospital (Unknown); The Third People's Hospital of Cangnan County (Unknown); Cangnan County Hospital of Traditional Chinese Medicine (Unknown); Pingyang County People's Hospital (Unknown); Pingyang County Hospital of Traditional Chinese Medicine (Unknown); Taishun County People's Hospital (Unknown); Taishun County Hospital of Traditional Chinese Medicine (Unknown); Yongjia County People's Medical Hospital (Unknown); Yongjia County Hospital of Traditional Chinese Medicine (Unknown); Wencheng County People's Hospital (Unknown); Shanghai Zhongshan Hospital (Other); Zhoushan Traditional Chinese Medicine Hospital (Unknown); Central Hospital of Dinghai District, Zhoushan City (Unknown); Putuo Hospital (Unknown); The First People's Hospital of Daishan County (Unknown); Shengsi County People's Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020-292
Record Dates: First submitted 2021-05-29; First posted 2021-06-07 (Actual); Last update posted 2021-07-22 (Actual); Status verified 2020-03

CONDITIONS: COVID-19 Pneumonia
Keywords: Emergency department; COVID-19; Epidemic prevention and control; Zhejiang province
MeSH Terms: conditions — Emergencies; COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The epidemic caused by the new coronavirus appeared in December 2019 and spread rapidly, and it has had a serious impact on the social development and people's lives in the world. On February 11, 2020, the World Health Organization (WHO) named the infectious disease caused by the virus COVID-19. my country classifies it as a Class B infectious disease, and controls it as a Class A infectious disease. In order to effectively respond to the epidemic, on January 23, 2020, Zhejiang Province first launched a first-level response to major public health emergencies across the country. Some patients with new coronary pneumonia, especially critically ill patients, may go to the emergency department first. Emergency medical staff must identify and isolate patients with new coronary pneumonia in a timely manner while ensuring the treatment of critically ill patients. People face greater unknowns and challenges in the anti-epidemic work. this research Participating in the prevention and control of the new crown pneumonia epidemic through investigations in the emergency department of Zhejiang Province Related conditions, to further improve the hospital's emergency medical service capabilities for reference.

DETAILED DESCRIPTION:
References：

1. Huang CL, Wang YM, Li XW, et al. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China[J]. Lancet, 2020, 395(10223): 497-506. DOI:10.1016/s0140-6736(20)30183-5.
2. Zhu N, Zhang DY, Wang WL, et al. A novel coronavirus from patients with pneumonia in China, 2019[J]. N Engl J Med, 2020, 382(8): 727- 733. DOI:10.1056/nejmoa2001017.
3. Gupta M, Abdelmaksoud A, Jafferany M, et al. COVID-19 and economy[J]. Dermatol Ther, 2020: e13329. DOI:10.1111/dth.13329.
4. Coronaviridae Study Group of the International Committee on Taxonomy of Viruses. The species severe acute respiratory syndrome- related coronavirus: classifying 2019-nCoV and naming it SARS- CoV-2 [J]. Nat Microbiol, 2020, 5(4):536-544. DOI:10.1038/s41564- 020-0695-z.
5. Lai CC, Shih TP, Ko WC, et al. Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) and coronavirus disease-2019 (COVID-19): The epidemic and the challenges[J]. Int J Antimicrob Agents, 2020, 55(3): 105924. DOI:10.1016/j.ijantimicag.2020.105924.

ELIGIBILITY:
Inclusion Criteria:

* County-level people's hospitals, TCM hospitals and above comprehensive public hospitals in Zhejiang Province;
* Voluntary participation in this study.

Exclusion Criteria:

* Incomplete data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Not applicable, not included in patients
Sampling Method: Non-Probability Sample
Enrollment: 181 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Basic information of the hospital | 7 day
  Hospital level, whether it is a designated hospital for COVID-19, whether it is capable of detecting nucleic acid for the new coronavirus, whether it has a fever clinic
Participation of the emergency department in fever clinics | 7 day
  The department/department responsible for the management of the fever clinic, whether the medical staff of the fever clinic has a fixed establishment, and the medical staff that temporarily supports the fever clinic source department
Patients with COVID-19 admitted to the emergency department | 7 day
  Number and distribution of patients
The frontline situation of emergency medical care support in the fight against the epidemic | 7 day
  Support the fever clinic of this hospital, isolation observation ward/confirmed ward, participate in the prehospital/inter-hospital transfer of new crown cases, participate in the hospital/regional prevention and management expert group, support the ward/ICU of designated hospitals in the province, support the ward of Hubei Province /ICU/ Fangcang shelter hospital
Epidemic prevention facilities in the emergency department | 7 day
  Number of spare separate consultation rooms, ordinary rescue rooms, and negative pressure rescue rooms, the supply of early anti-epidemic protective equipment

CONTACTS AND LOCATIONS:
Overall Officials: Mao Zhang, MD, Study Chair — Second Affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital, Zhejiang University School of Medicine & Institute of Emergency Medicine, Zhejiang University, Hangzhou, Zhejiang, China